CLINICAL TRIAL: NCT03835533
Title: A Multicenter, Open-Label, Exploratory Platform Study to Evaluate Biomarkers and Immunotherapy Combinations for the Treatment of Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: Platform Study for Prostate Researching Translational Endpoints Correlated to Response to Inform Use of Novel Combinations
Acronym: PORTER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parker Institute for Cancer Immunotherapy (Other)
Collaborators: Bristol-Myers Squibb (Industry); Celldex Therapeutics (Industry); Cancer Research Institute, New York City (Other); Inovio Pharmaceuticals (Industry); Oncovir, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PICI0033
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: Metastatic Castration-resistant Prostate Cancer; Immunotherapy; Platform study; NKTR-214; Nivolumab; CDX-301; Poly-ICLC; INO-5151
MeSH Terms: interventions — bempegaldesleukin; Nivolumab; Radiosurgery; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: NKTR-214 + Nivolumab (Experimental)
  Interventions: Drug: NKTR-214 (Cohort A); Drug: Nivolumab (Cohort A, B and C)
- Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab (Experimental)
  Interventions: Drug: Nivolumab (Cohort A, B and C); Radiation: Stereotactic body radiation therapy (SBRT) (Cohort B); Drug: CDX-301 (Cohort B and C); Drug: Poly-ICLC (Cohort B)
- Cohort C: CDX-301 + INO-5151 + Nivolumab (Experimental)
  Interventions: Drug: Nivolumab (Cohort A, B and C); Drug: CDX-301 (Cohort B and C); Drug: INO-5151 (Cohort C); Device: Cellectra 2000

INTERVENTIONS:
Drug: NKTR-214 (Cohort A) — NKTR-214 will be administered intravenously every 3 weeks for up to 2 years
  Arms: Cohort A: NKTR-214 + Nivolumab
Drug: Nivolumab (Cohort A, B and C) — Nivolumab will be administered intravenously every 3 weeks for up to 2 years to cohort A, every 4 weeks for up to 2 years for cohort B and C.
  Other Names: Opdivo
Radiation: Stereotactic body radiation therapy (SBRT) (Cohort B) — Radiation therapy will be administered at 30 - 50 Gy in 1 - 5 doses, starting on Day 1 or 2 of Cycle 1
  Arms: Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab
Drug: CDX-301 (Cohort B and C) — CDX-301 will be subcutaneously once a day for 5 days for cohort B. CDX-301 will be subcutaneously once a day for 10 days of immune-priming lead-in for cohort C.
  Arms: Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab; Cohort C: CDX-301 + INO-5151 + Nivolumab
Drug: Poly-ICLC (Cohort B) — Poly-ICLC will be administered intramuscularly twice weekly for 3 weeks starting on Day 1 of Cycle 1
  Arms: Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab
Drug: INO-5151 (Cohort C) — INO-5151 will be administered intramuscularly on Day 8 of the Immune-priming Lead-in, and on day 1 of Cycle 1, 2 and 3, then every 12 weeks thereafter
  Arms: Cohort C: CDX-301 + INO-5151 + Nivolumab
Device: Cellectra 2000 — Electroporation device
  Arms: Cohort C: CDX-301 + INO-5151 + Nivolumab

SUMMARY:
This study is designed to evaluate multiple clinical hypotheses and mechanistically-defined combinations to evaluate the safety and efficacy of immunotherapy combinations in participants with mCRPC who have received prior secondary androgen receptor signaling inhibitor therapy (eg, abiraterone, enzalutamide, apalutamide).

DETAILED DESCRIPTION:
This is an open-label, non-randomized, exploratory platform protocol designed to assess the safety and antitumor activity of multiple immunotherapy combinations in participants with mCRPC who have received prior therapy. The platform study will consist of 2 stages: Stage 1, an initial stage to evaluate safety, biomarkers, and clinical activity of a combination and Stage 2, an expanded cohort, when warranted, based on the safety, clinical activity, and/or biomarker results from Stage 1. The Sponsor intends to modify and/or add new combinations to the protocol as data emerge from this and other trials.

Participants must provide consent for archival tissue from a prior biopsy or surgery for prostate cancer and must consent to baseline and on-treatment biopsies, if medically feasible. Participants will be assigned to receive one of the enrolling combination study interventions and will be monitored for safety and response.

ELIGIBILITY:
Key Inclusion Criteria:

1. Metastatic castration resistant prostate cancer with castrate-level testosterone (< 50 ng/dL) at screening.
2. Disease progression per Prostate Cancer Working Group 3 (PCWG3) criteria.
3. Provide fresh pre-treatment core needle or incisional biopsy of a metastatic tumor lesion not previously irradiated. Fine needle aspiration is not acceptable.

   1. Additionally, if a pre-treatment biopsy is not medically feasible for participants with bone only disease, formalin-fixed paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or at least 10 slides containing unstained, freshly cut, serial sections must be provided.
   2. For all participants, in addition to fresh pre-treatment biopsy, consent for archival tissue is required.
4. Must be willing to undergo tumor biopsy(ies) on treatment, if medically feasible.
5. Have received and progressed on prior secondary androgen receptor signaling inhibitor therapy (eg, abiraterone, enzalutamide, apalutamide).
6. Participants must discontinue antiandrogen therapy (ie, bicalutamide, flutamide, nilutamide) at least 4-6 weeks prior to registration with no evidence of prostate-specific antigen (PSA) decline after washout.

   1. Bicalutamide: Washout period at least 6 weeks
   2. Flutamide and nilutamide: Washout period at least 4 weeks
7. Participants must discontinue therapies for mCRPC for 5 half-lives or 28 days, whichever is shorter.

   1. Participants will remain on gonadotropin-releasing hormone (GnRH) agents throughout this study.
   2. Prior chemotherapy is allowed if no progression of disease on chemotherapy as defined by PCWG3-modified RECIST 1.1.
   3. Prior treatment with sipuleucel-T, radium-223, or poly ADP ribose polymerase (PARP) inhibitor (eg, olaparib) is allowed.
   4. Tissue biopsy may be performed during washout period.

Key Exclusion Criteria:

1. Has a diagnosis of immunodeficiency or conditions that need systemic corticosteroid replacement therapy > 10 mg/day prednisone (or equivalent) or other immunosuppressive medications within 28 days prior to the first dose of study intervention. Inhaled steroids are permitted if necessary.
2. Has any active known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, controlled autoimmune hypothyroidism, psoriasis not requiring systemic treatment, or other conditions under control are permitted to enroll.
3. Has a known history of active TB (Bacillus Tuberculosis).
4. Has known history of, or any evidence of active, non-infectious pneumonitis.
5. Known history of testing positive for human immunodeficiency virus (HIV), known acquired immunodeficiency syndrome (AIDS), or any positive test for hepatitis B or hepatitis C virus representing acute or chronic disease.
6. Has received a live vaccine within 30 days of planned start of study intervention.

   Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (eg, Flu-Mist®) are live attenuated vaccines, and are not allowed.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of study intervention and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study intervention. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-06-21 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parker Institute for Cancer Immunotherapy, Study Director — Parker Institute for Cancer Immunotherapy
Locations (6):
- United States (6):
  - Angeles Clinic, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Beer TM, Kwon ED, Drake CG, Fizazi K, Logothetis C, Gravis G, Ganju V, Polikoff J, Saad F, Humanski P, Piulats JM, Gonzalez Mella P, Ng SS, Jaeger D, Parnis FX, Franke FA, Puente J, Carvajal R, Sengelov L, McHenry MB, Varma A, van den Eertwegh AJ, Gerritsen W. Randomized, Double-Blind, Phase III Trial of Ipilimumab Versus Placebo in Asymptomatic or Minimally Symptomatic Patients With Metastatic Chemotherapy-Naive Castration-Resistant Prostate Cancer. J Clin Oncol. 2017 Jan;35(1):40-47. doi: 10.1200/JCO.2016.69.1584. Epub 2016 Oct 31. PMID 28034081
- [Background] Di Lorenzo G, Buonerba C, Kantoff PW. Immunotherapy for the treatment of prostate cancer. Nat Rev Clin Oncol. 2011 May 24;8(9):551-61. doi: 10.1038/nrclinonc.2011.72. PMID 21606971
- [Background] Drake CG. Prostate cancer as a model for tumour immunotherapy. Nat Rev Immunol. 2010 Aug;10(8):580-93. doi: 10.1038/nri2817. PMID 20651745
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Flammiger A, Bayer F, Cirugeda-Kuhnert A, Huland H, Tennstedt P, Simon R, Minner S, Bokemeyer C, Sauter G, Schlomm T, Trepel M. Intratumoral T but not B lymphocytes are related to clinical outcome in prostate cancer. APMIS. 2012 Nov;120(11):901-8. doi: 10.1111/j.1600-0463.2012.02924.x. Epub 2012 Jul 4. PMID 23009114
- [Background] Gao J, Ward JF, Pettaway CA, Shi LZ, Subudhi SK, Vence LM, Zhao H, Chen J, Chen H, Efstathiou E, Troncoso P, Allison JP, Logothetis CJ, Wistuba II, Sepulveda MA, Sun J, Wargo J, Blando J, Sharma P. VISTA is an inhibitory immune checkpoint that is increased after ipilimumab therapy in patients with prostate cancer. Nat Med. 2017 May;23(5):551-555. doi: 10.1038/nm.4308. Epub 2017 Mar 27. PMID 28346412
- [Background] Graff JN, Alumkal JJ, Drake CG, Thomas GV, Redmond WL, Farhad M, Cetnar JP, Ey FS, Bergan RC, Slottke R, Beer TM. Early evidence of anti-PD-1 activity in enzalutamide-resistant prostate cancer. Oncotarget. 2016 Aug 16;7(33):52810-52817. doi: 10.18632/oncotarget.10547. PMID 27429197
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Kwon ED, Drake CG, Scher HI, Fizazi K, Bossi A, van den Eertwegh AJ, Krainer M, Houede N, Santos R, Mahammedi H, Ng S, Maio M, Franke FA, Sundar S, Agarwal N, Bergman AM, Ciuleanu TE, Korbenfeld E, Sengelov L, Hansen S, Logothetis C, Beer TM, McHenry MB, Gagnier P, Liu D, Gerritsen WR; CA184-043 Investigators. Ipilimumab versus placebo after radiotherapy in patients with metastatic castration-resistant prostate cancer that had progressed after docetaxel chemotherapy (CA184-043): a multicentre, randomised, double-blind, phase 3 trial. Lancet Oncol. 2014 Jun;15(7):700-12. doi: 10.1016/S1470-2045(14)70189-5. Epub 2014 May 13. PMID 24831977
- [Background] Lee P, Gujar S. Potentiating prostate cancer immunotherapy with oncolytic viruses. Nat Rev Urol. 2018 Apr;15(4):235-250. doi: 10.1038/nrurol.2018.10. Epub 2018 Feb 13. PMID 29434366
- [Background] Lopez-Bujanda Z, Drake CG. Myeloid-derived cells in prostate cancer progression: phenotype and prospective therapies. J Leukoc Biol. 2017 Aug;102(2):393-406. doi: 10.1189/jlb.5VMR1116-491RR. Epub 2017 May 26. PMID 28550116
- [Background] Martin AM, Nirschl TR, Nirschl CJ, Francica BJ, Kochel CM, van Bokhoven A, Meeker AK, Lucia MS, Anders RA, DeMarzo AM, Drake CG. Paucity of PD-L1 expression in prostate cancer: innate and adaptive immune resistance. Prostate Cancer Prostatic Dis. 2015 Dec;18(4):325-32. doi: 10.1038/pcan.2015.39. Epub 2015 Aug 11. PMID 26260996
- [Background] McNeel DG, Bander NH, Beer TM, Drake CG, Fong L, Harrelson S, Kantoff PW, Madan RA, Oh WK, Peace DJ, Petrylak DP, Porterfield H, Sartor O, Shore ND, Slovin SF, Stein MN, Vieweg J, Gulley JL. The Society for Immunotherapy of Cancer consensus statement on immunotherapy for the treatment of prostate carcinoma. J Immunother Cancer. 2016 Dec 20;4:92. doi: 10.1186/s40425-016-0198-x. eCollection 2016. PMID 28031820
- [Background] Miller AM, Lundberg K, Ozenci V, Banham AH, Hellstrom M, Egevad L, Pisa P. CD4+CD25high T cells are enriched in the tumor and peripheral blood of prostate cancer patients. J Immunol. 2006 Nov 15;177(10):7398-405. doi: 10.4049/jimmunol.177.10.7398. PMID 17082659
- [Background] Pasero C, Gravis G, Guerin M, Granjeaud S, Thomassin-Piana J, Rocchi P, Paciencia-Gros M, Poizat F, Bentobji M, Azario-Cheillan F, Walz J, Salem N, Brunelle S, Moretta A, Olive D. Inherent and Tumor-Driven Immune Tolerance in the Prostate Microenvironment Impairs Natural Killer Cell Antitumor Activity. Cancer Res. 2016 Apr 15;76(8):2153-65. doi: 10.1158/0008-5472.CAN-15-1965. Epub 2016 Apr 5. PMID 27197252
- [Background] Patel A, Fong L. Immunotherapy for Prostate Cancer: Where Do We Go From Here?-PART 1: Prostate Cancer Vaccines. Oncology (Williston Park). 2018 Mar 15;32(3):112-20. PMID 29548065
- [Background] Redman JM, Steinberg SM, Gulley JL. Quick efficacy seeking trial (QuEST1): a novel combination immunotherapy study designed for rapid clinical signal assessment metastatic castration-resistant prostate cancer. J Immunother Cancer. 2018 Sep 18;6(1):91. doi: 10.1186/s40425-018-0409-8. PMID 30227893
- [Background] Scher HI, Halabi S, Tannock I, Morris M, Sternberg CN, Carducci MA, Eisenberger MA, Higano C, Bubley GJ, Dreicer R, Petrylak D, Kantoff P, Basch E, Kelly WK, Figg WD, Small EJ, Beer TM, Wilding G, Martin A, Hussain M; Prostate Cancer Clinical Trials Working Group. Design and end points of clinical trials for patients with progressive prostate cancer and castrate levels of testosterone: recommendations of the Prostate Cancer Clinical Trials Working Group. J Clin Oncol. 2008 Mar 1;26(7):1148-59. doi: 10.1200/JCO.2007.12.4487. PMID 18309951
- [Background] Scher HI, Morris MJ, Stadler WM, Higano C, Basch E, Fizazi K, Antonarakis ES, Beer TM, Carducci MA, Chi KN, Corn PG, de Bono JS, Dreicer R, George DJ, Heath EI, Hussain M, Kelly WK, Liu G, Logothetis C, Nanus D, Stein MN, Rathkopf DE, Slovin SF, Ryan CJ, Sartor O, Small EJ, Smith MR, Sternberg CN, Taplin ME, Wilding G, Nelson PS, Schwartz LH, Halabi S, Kantoff PW, Armstrong AJ; Prostate Cancer Clinical Trials Working Group 3. Trial Design and Objectives for Castration-Resistant Prostate Cancer: Updated Recommendations From the Prostate Cancer Clinical Trials Working Group 3. J Clin Oncol. 2016 Apr 20;34(12):1402-18. doi: 10.1200/JCO.2015.64.2702. Epub 2016 Feb 22. PMID 26903579
- [Background] Sydes MR, Spears MR, Mason MD, Clarke NW, Dearnaley DP, de Bono JS, Attard G, Chowdhury S, Cross W, Gillessen S, Malik ZI, Jones R, Parker CC, Ritchie AWS, Russell JM, Millman R, Matheson D, Amos C, Gilson C, Birtle A, Brock S, Capaldi L, Chakraborti P, Choudhury A, Evans L, Ford D, Gale J, Gibbs S, Gilbert DC, Hughes R, McLaren D, Lester JF, Nikapota A, O'Sullivan J, Parikh O, Peedell C, Protheroe A, Rudman SM, Shaffer R, Sheehan D, Simms M, Srihari N, Strebel R, Sundar S, Tolan S, Tsang D, Varughese M, Wagstaff J, Parmar MKB, James ND; STAMPEDE Investigators. Adding abiraterone or docetaxel to long-term hormone therapy for prostate cancer: directly randomised data from the STAMPEDE multi-arm, multi-stage platform protocol. Ann Oncol. 2018 May 1;29(5):1235-1248. doi: 10.1093/annonc/mdy072. PMID 29529169
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Wolchok JD, Hoos A, O'Day S, Weber JS, Hamid O, Lebbe C, Maio M, Binder M, Bohnsack O, Nichol G, Humphrey R, Hodi FS. Guidelines for the evaluation of immune therapy activity in solid tumors: immune-related response criteria. Clin Cancer Res. 2009 Dec 1;15(23):7412-20. doi: 10.1158/1078-0432.CCR-09-1624. Epub 2009 Nov 24. PMID 19934295

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
Started | 14 | 15 | 14
Completed | 6 | 3 | 3
Not Completed | 8 | 12 | 11
Not completed — Death | 5 | 10 | 9
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab | Total
Number analyzed (Participants) | 14 | 15 | 14 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 4 | 19
  >=65 years | 5 | 9 | 10 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (6.9) | 69.7 (10.3) | 71.4 (9.3) | 68.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 14 | 15 | 14 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 2 | 7
  Not Hispanic or Latino | 14 | 10 | 12 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 2 | 0 | 0 | 2
  Race: Black or African American | 0 | 3 | 2 | 5
  Race: White | 12 | 8 | 11 | 31
  Race: Other | 0 | 4 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 15 | 14 | 43
ECOG Performance Score at Screening [Count of Participants; unit: Participants] — Measure Description: The ECOG (Eastern Cooperative Oncology Group) performance status is a widely-used scale to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine the appropriate treatment and prognosis.
  Here is a brief description of the ECOG performance status:
  0: Fully active, able to carry on all pre-disease performance without restriction.
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework or office work.
  Participants
    0 | 8 | 8 | 10 | 26
    1 | 5 | 7 | 4 | 16
    Missing | 1 | 0 | 0 | 1
Cancer Stage at Initial Diagnosis [Count of Participants; unit: Participants] — The stage of cancer at initial diagnosis provides vital information about the extent of cancer in the body and is pivotal for prognosis and treatment decisions. Cancer stages typically range from stage 0 (in situ, localized growth) to stage 4 (advanced cancer with distant metastasis).
  Participants
    Stage 1 | 2 | 1 | 0 | 3
    Stage 2 | 2 | 2 | 1 | 5
    Stage 3 | 2 | 2 | 4 | 8
    Stage 4 | 8 | 8 | 8 | 24
    Unknown | 0 | 2 | 1 | 3
Prostate-Specific Antigen (PSA) (ng/mL) at Baseline [Median (Full Range); unit: ng/mL] | 25.3 [0.2 to 97.9] | 37.1 [1.3 to 2651.0] | 43.0 [3.5 to 3945.5] | 32.7 [0.2 to 3945.5]
Circulating Tumor Cells (CTC) value (cells/7.5 mL of blood) at Baseline [Median (Full Range); unit: cells/7.5 mL of blood] — Population: Patients were excluded from the calculation if there was not a sufficient quantity of blood in the patient's collection tube to obtain a result.
  cells/7.5 mL of blood
    number analyzed (Participants) | 10 | 13 | 14 | 37
    (all) | 4.5 [0 to 1934] | 13.0 [0 to 150] | 5.5 [0 to 60] | 5.0 [0 to 1934]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE is any event that either occurs after the initiation of study drug, having been absent at baseline, or, if present at baseline, appears to have worsened in severity or frequency, regardless of its relation to the drug. An SAE is any AE that suggests a significant hazard, contraindication, side effect, or untoward medical occurrence that results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
  Investigators recorded AEs during each participant interaction. Prior to initiation of study drug, only SAEs that were related to a protocol-mandated intervention were recorded.
  The AE row includes all participants who experienced at least one AE, including SAEs.
Time Frame: For AEs, from initiation of study drug through 100 days after last dose, up to 24 months. For SAEs, from signing informed consent (prior to Screening) through 100 days after last dose, up to 24 months.
Population: The evaluable population is defined as all participants in a cohort who received at least one dose of any component of the combination study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
Number analyzed (Participants) | 14 | 15 | 14
Participants
  Adverse Events (AEs) | 14 | 15 | 13
  Serious Adverse Events (SAEs) | 7 | 4 | 5

2. Secondary Outcome: Composite Response Rate (CRR)
Description: CRR is a composite endpoint where response is defined as a participant meeting at least one of the following:
  1. circulating tumor cells (CTC) change from unfavorable (≥ 5 cells/7.5 mL of blood) to favorable (<= 4 cells/7.5 mL of blood);
  2. ≥ 50% reduction in Prostate-Specific Antigen (PSA) from baseline, with a repeat assessment confirming the results at least 3 weeks later;
  3. Per Prostate Cancer Clinical Trials Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, a complete response (CR; disappearance of all target and non-target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions). A repeat tumor assessment must confirm the CR/PR results at least 3 weeks later.
Time Frame: Initiation of study drug through radiographic progression or initiation of new anti-cancer therapy, whichever occurred first, up to 20 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
Number analyzed (Participants) | 14 | 15 | 14
Participants | 1 | 5 | 1

3. Secondary Outcome: Disease Control Rate (DCR)
Description: Per Prostate Cancer Clinical Trials Working Group 3 (PCWG3)-modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, a complete response (CR) is defined as disappearance of all target and non-target lesions and a partial response (PR) as a >=30% decrease in the sum of the longest diameter of target lesions. A repeat tumor assessment must confirm the CR/PR results at least 3 weeks later. DCR = CR + PR + stable disease lasting at least 6 months.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
Number analyzed (Participants) | 14 | 15 | 14
Participants | 2 | 5 | 2

4. Secondary Outcome: Radiographic Progression-free Survival (rPFS)
Description: Defined as time from initiation of study intervention to the first objective evidence of radiographic progression, or death due to any cause (whichever occurs first). Per Prostate Cancer Clinical Trials Working Group 3 (PCWG3)-modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST) version 1.1, radiographic progression is defined using as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new non-bone lesions, or at least 2 new bone lesions relative to the first post-treatment scan that are confirmed on a subsequent scan.
  rPFS and confidence intervals were estimated using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
Number analyzed (Participants) | 14 | 15 | 14
months | 2.8 [2.00 to 7.26] | 7.5 [3.52 to 10.48] | 3.2 [2.66 to 10.28]

5. Secondary Outcome: Overall Survival (OS)
Description: Defined as the time from initiation of study invention until death due to any cause. OS and confidence intervals were estimated using the Kaplan-Meier method.
Time Frame: From initiation of study drug until death due to any cause, up to 2.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
Number analyzed (Participants) | 14 | 15 | 14
months | NA [9.04 to NA] — The median and upper confidence limit is not estimable due to an insufficient number of participants with an event | 20.6 [5.65 to 27.50] | 17.3 [3.48 to NA] — The median and upper confidence limit is not estimable due to an insufficient number of participants with an event

6. Secondary Outcome: Overall Survival (OS) at 12 Months
Description: Defined as the overall survival probability at 12 months, calculated using the Kaplan-Meier method.
Time Frame: At 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
Number analyzed (Participants) | 14 | 15 | 14
probability | 0.579 [0.260 to 0.801] | 0.525 [0.252 to 0.740] | 0.524 [0.227 to 0.754]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from initiation of study drug through 100 days after last dose, up to 24 months. Serious adverse events (SAEs) were collected from signing informed consent (prior to Screening) through 100 days after last dose, up to 24 months. All-cause mortality was collected from initiation of study drug, up to 2.5 years.
Description: Investigators recorded AEs during each participant interaction. Prior to initiation of study drug, only SAEs that were related to a protocol-mandated intervention were recorded.
Arm/Group | Cohort A: NKTR-214 + Nivolumab | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab | Cohort C: CDX-301 + INO-5151 + Nivolumab
All-Cause Mortality (participants affected / at risk) | 5/14 | 10/15 | 9/14
Serious Adverse Events (participants affected / at risk) | 7/14 | 4/15 | 5/14
Other Adverse Events (participants affected / at risk) | 13/14 | 15/15 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: NKTR-214 + Nivolumab (N=14) | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab (N=15) | Cohort C: CDX-301 + INO-5151 + Nivolumab (N=14)
Endocarditis (Infections and infestations) | 2 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: NKTR-214 + Nivolumab (N=14) | Cohort B: SBRT + CDX-301 + Poly-ICLC + Nivolumab (N=15) | Cohort C: CDX-301 + INO-5151 + Nivolumab (N=14)
Fatigue (General disorders) | 6 | 2 | 5
Pyrexia (General disorders) | 6 | 1 | 0
Chills (General disorders) | 4 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 1
Influenza like illness (General disorders) | 1 | 1 | 0
Injection site reaction (General disorders) | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 1 | 0 | 0
Injection site discomfort (General disorders) | 0 | 0 | 1
Injection site irritation (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Tenderness (General disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Autoimmune arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 1
Nausea (Gastrointestinal disorders) | 3 | 4 | 2
Constipation (Gastrointestinal disorders) | 1 | 4 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 4 | 2
Alanine aminotransferase increased (Investigations) | 4 | 2 | 2
Blood creatinine increased (Investigations) | 4 | 2 | 0
Lymphocyte count decreased (Investigations) | 5 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 2
Weight decreased (Investigations) | 1 | 2 | 1
White blood cell count decreased (Investigations) | 2 | 2 | 0
Platelet count decreased (Investigations) | 2 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0
Troponin I increased (Investigations) | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 4
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 3
Cognitive disorder (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 2
Flushing (Vascular disorders) | 3 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1
Hot flush (Vascular disorders) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 0 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 4 | 2 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Haemoglobinuria (Renal and urinary disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1
Eyelid function disorder (Eye disorders) | 1 | 0 | 0
Hypermetropia (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial Site and/or Co-Principal Investigators may publish or present Study Data and other results of the Study from the Trial Site individually upon the first to occur of: (i) twelve (12) months after conclusion, abandonment, or termination of the Study at all Affiliated Research Institutions, or (ii) after Parker Institute for Cancer Immunotherapy [PICI] confirms in writing there will not be a multi-site Study publication.

DOCUMENTS (5):
  • Study Protocol: Cohort A (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT03835533/Prot_000.pdf
  • Study Protocol: Cohort B (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT03835533/Prot_001.pdf
  • Study Protocol: Cohort C (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03835533/Prot_002.pdf
  • Study Protocol: Core protocol (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT03835533/Prot_003.pdf
  • Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT03835533/SAP_004.pdf